CLINICAL TRIAL: NCT02338219
Title: Effects of Pregnancy and Childbirth on Pelvic Floor Morphology and Sexual Function in Egyptian Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, al-azhar unversity (assuit), faculty of medicine, obstetrics and gynecology department, Al-Azhar University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U1111-1159-6256
Record Dates: First submitted 2014-08-22; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Pregnancy, Childbirth and Puerperal Disorders
Keywords: postpartum pelvic floor
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- vaginal delivery (Active Comparator): postpartum female pelvic floor muscle affection postpartum sexual function in Egyptian women.
  Interventions: Other: postpartum female pelvic floor muscle affection; Other: postpartum sexual function in Egyptian women.
- elective cesarean section (Active Comparator): postpartum female pelvic floor muscle affection postpartum sexual function in Egyptian women.
  Interventions: Other: postpartum female pelvic floor muscle affection; Other: postpartum sexual function in Egyptian women.
- urgent cesarean section (Active Comparator): postpartum female pelvic floor muscle affection postpartum sexual function in Egyptian women.
  Interventions: Other: postpartum female pelvic floor muscle affection

INTERVENTIONS:
Other: postpartum female pelvic floor muscle affection — transperineal pelvic floor ultrasound applied for the submitted 120 women "primiparae" (40 women after normal vaginal delivery), (40 women after urgent cesarean section), (40 women after elective cesarean section), in early postpartum period (48 to 72) hours postpartum, to evaluate levator ani morphology.
Other: postpartum sexual function in Egyptian women. — answering of the validated female sexual function index (F.S.F.I) three months postpartum period for same cases submitted to ultrasound.
  Arms: elective cesarean section; vaginal delivery

SUMMARY:
The purpose of this study is t o evaluate levator ani morphology following normal vaginal delivery and cesarean section (elective and emergent), using three-dimensional (3D) ultrasound, and to study the effect of mode of delivery on female sexual function.

DETAILED DESCRIPTION:
1. transperineal pelvic floor ultrasound applied for the submitted 120 women "primiparae" (40 women after normal vaginal delivery), (40 women after urgent cesarean section), (40 women after elective cesarean section), in early postpartum period (48 to 72) hours postpartum, to evaluate levator ani morphology.
2. answering of the validated female sexual function index (F.S.F.I) three months postpartum period for same cases submitted to ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* primiparae in early postpartum period (48 hours to72 hours). written consent was taken. easy communicable, reachable women for further requirements.

Exclusion Criteria:

* Refused consent. 2. Previous vaginal or cesarean delivery. 3. Severe mental illness. 4. Severe physical handicap or difficulties in communication. 5. Women without postpartum active sexual life or separate from their spouse. 6. Past history of sexual dysfunction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength as assessed by three/four dimensional translabial pelvic floor ultrasound had worst morbidity after normal vaginal delivery | early postpartum period (48 to 72) hours postpartum

SECONDARY OUTCOMES:
Sexual function of pelvic floor as assessed by the validated female sexual function index questionnaire was impaired in all women after delivery | at 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, prof, Principal Investigator — Al-Azhar University; Muhamed Osman Osman, Study Chair — Al-Azhar University